CLINICAL TRIAL: NCT05017116
Title: A Single and Repeated Dose Escalation, Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics and Preliminary Pharmacodynamics of RBD1016 in Subjects with Chronic Hepatitis B Virus (HBV) Infection
Brief Title: A Single and Repeated Dose Escalation of RBD1016 in Subjects with Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBHB1103-HK
Record Dates: First submitted 2021-08-10; First posted 2021-08-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-10

CONDITIONS: Chronic Hepatitis B
Keywords: CHB; chronic hepatitis B infection
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A，single dose group (Experimental): Subjects will receive single dose RBD1016/placebo on D1 combined with antiviral drugs during the study period.
  Interventions: Drug: RBD1016; Drug: Placebo; Drug: Entecavir
- Part B, multiple dose group (Experimental): Subjects will receive two doses of RBD1016/placebo on D1 and D29 combined with antiviral drugs during the study period.
  Interventions: Drug: RBD1016; Drug: Placebo; Drug: Entecavir

INTERVENTIONS:
Drug: RBD1016 — subcutaneous injection
  Other Names: RBD1016 injection
Drug: Placebo — subcutaneous injection
Drug: Entecavir — Take orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single (Part A) and repeated dose (Part B) escalation, phase I clinical study to evaluate the safety, pharmacokinetics (PK) and preliminary pharmacodynamics (PD) of RBD1016 in subjects with chronic HBV infection.

DETAILED DESCRIPTION:
The study consists of two parts. Part A is the single dose escalation study where subjects with chronic HBV infection will be assigned to receive single dose of RBD1016 or placebo . Part B is the multiple dose escalation study where subjects with chronic HBV infection will be assigned to receive two doses of RBD1016 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in this clinical trial, are able to correctly understand and have signed the informed consent in writing;
2. Male or female volunteer aged 18-55 years (inclusive);
3. Body Mass Index (BMI) of 18-30 kg/m2 (inclusive);
4. Subjects with chronic HBV infection, including immunotolerant subjects, treatment naïve subjects and treated subjects.
5. Ability to cooperate with study staff and comply with the study requirements and follow the protocol-specified procedures.

Exclusion Criteria:

1. Subjects with liver diseases other than hepatitis B, including hepatitis C, hemochromatosis, primary sclerosing cholangitis; alcoholic, drug-related or autoimmune liver diseases; primary liver cancer and indeterminate nodules on liver imaging test;
2. A history or manifestations of liver decompensation (e.g. Child-Pugh Class B or C, or ascites, gastrointestinal bleeding, hepatic encephalopathy or spontaneous bacterial peritonitis, etc.);
3. Transient elastography at screening revealing FibroScan value ≥ 9 kPa or liver biopsy evidencing hepatic fibrosis within 24 months;
4. The following laboratory findings: total serum bilirubin> 2×ULN; serum alpha-fetoprotein>50μg/L; serum albumin <3.5g/dL; international normalized ratio (INR)> 1.25; serum creatinine > 1.5×ULN; any laboratory outliers of clinical significance that in the investigator's opinion may interfere with the interpretation of efficacy or safety data;
5. 12-lead ECG abnormalities with clinical significance;
6. Pregnant or lactating women or women of child-bearing potential who are unwilling to take effective contraception throughout the course of the study (refer to Appendix 3 for details);
7. Other factors that in the investigator's opinion would make it inappropriate for the subject to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) within 28 days after treatment (Part A) | up to 28 days
  All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).AEs and SAEs occurred throughout the course of the study will be evaluated and graded based on NCI-CTCAE V5.0.
Adverse events (AEs) and serious adverse events (SAEs) within 28 days after the last treatment(Part B) | up to 28 days
  All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).AEs and SAEs occurred throughout the course of the study will be evaluated and graded based on NCI-CTCAE V5.0.

SECONDARY OUTCOMES:
To draw the figure of HBsAg dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B surface antigen (HBsAg).
To draw the figure of HBsAb dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B surface antibody (HBsAb).
To draw the figure of HBeAg dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B e antigen (HBeAg).
To draw the figure of HBeAb dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B e antibody (HBeAb).
To draw the figure of HBcAb dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B core antibody (HBcAb).
To draw the figure of HBcrAg dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B core-related antigen (HBcrAg).
To draw the figure of HBV DNA dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  PCR will be used to detect HBV DNA.
To draw the figure of HBV RNA dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  PCR will be used to detect HBV RNA.
To draw the figure of peripheral blood T lymphocyte subsets dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Flow Cytometry will be used to detect peripheral blood T lymphocyte subsets.
To draw the figure of B cell dynamic changes from baseline to Week 24 (Part A). | up to 24 weeks
  Flow Cytometry will be used to detect B cell count.
To characterize the pharmacokinetic parameter Cmax (Part A). | up to 85 days
  PCR will be ued to detect Maximum concentration (Cmax) and PhoenixWinNonlin software (V8.0 or higher) will be used to calculate the PK parameters.
To characterize the pharmacokinetic parameter Tmax (Part A). | up to 85 days
  Time to maximum concentration (Tmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher) will be used to calculate the PK parameter.
To characterize the pharmacokinetic parameter AUC0-t (Part A). | up to 85 days
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter AUC0-inf (Part A). | up to 85 days
  Area under the concentration-time curve from 0 to infinity (AUC0-inf) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter t1/2 (Part A). | up to 85 days
  Half-Life (t1/2) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter Vd (Part A). | up to 85 days
  Apparent volume of distribution (Vd) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter CL/F (Part A) | up to 85 days
  Clearance (CL/F) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To draw the figure of HBsAg dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B surface antigen (HBsAg).
To draw the figure of HBsAb dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B surface antibody (HBsAb).
To draw the figure of HBeAg dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B e antigen (HBeAg).
To draw the figure of HBeAb dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B e antibody (HBeAb).
To draw the figure of HBcAb dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B core antibody (HBcAb).
To draw the figure of HBcrAg dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Electro chmiluminescence method will be used to detect hepatitis B core-related antigen (HBcrAg).
To draw the figure of HBV DNA dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  PCR will be used to detect HBV DNA.
To draw the figure of HBV RNA dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  PCR will be used to detect HBV RNA.
To draw the figure of peripheral blood T lymphocyte subsets dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Flow Cytometry will be used to detect peripheral blood T lymphocyte subsets.
To draw the figure of B cell dynamic changes from baseline to Week 24 (Part B). | up to 24 weeks
  Flow Cytometry will be used to detect B cell count.
To characterize the pharmacokinetic parameter Cmax (Part B). | up to 113 days
  PCR will be ued to detect Maximum concentration (Cmax) and PhoenixWinNonlin software (V8.0 or higher) will be used to calculate the PK parameters.
To characterize the pharmacokinetic parameter Tmax (Part B). | up to 113 days
  Time to maximum concentration (Tmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher) will be used to calculate the PK parameter.
To characterize the pharmacokinetic parameter AUC0-t (Part B). | up to 113 days
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter AUC0-inf (Part B). | up to 113 days
  Area under the concentration-time curve from 0 to infinity (AUC0-inf) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter t1/2 (Part B). | up to 113 days
  Half-Life (t1/2) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter Vd (Part B). | up to 113 days
  Apparent volume of distribution (Vd) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
To characterize the pharmacokinetic parameter CL/F (Part B). | up to 113 days
  Clearance (CL/F) will be calculated by PhoenixWinNonlin software (V8.0 or higher).

CONTACTS AND LOCATIONS:
Overall Officials: Walter Seto, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No